CLINICAL TRIAL: NCT01886781
Title: Randomised Controlled Trial: Effect of Lactobacillus Plantarum 299v on Symptoms of Irritable Bowel Syndrome
Brief Title: Effect of Lactobacillus Plantarum 299v on Symptoms of Irritable Bowel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Stellenbosch (Other)
Collaborators: Nestlè Nutrition Institute Africa (Other); National Research Foundation (NRF) (RSA) (Unknown)
Responsible Party: Principal Investigator, Cheryl Stevenson, Mrs, University of Stellenbosch
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N10-08-270
Record Dates: First submitted 2013-06-18; First posted 2013-06-26 (Estimated); Results first posted 2014-09-29 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-09

CONDITIONS: Irritable Bowel Syndrome
Keywords: only constipation and diarrhea predominant; no mixed or alternating types
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Jogging

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lactobacillus plantarum 299v (Experimental): Lactobacillus plantarum 299v capsules
  Interventions: Drug: Lactobacillus plantarum 299v; Other: Run in period; Other: Wash - out period
- Crytalline cellulose powder (Placebo Comparator): Placebo capsule, filled with micro-crystalline cellulose powder
  Interventions: Drug: Placebo comparator; Other: Run in period; Other: Wash - out period
- Run in period (No Intervention): Run in period of one to two weeks, no treatment. At baseline randomization and treatment commenced.
- Wash out period (No Intervention): Wash out period of two weeks, no treatment.

INTERVENTIONS:
Drug: Lactobacillus plantarum 299v — two capsules of 5 X 10 ^9 c.f.u each
  Other Names: Lp 299v
  Arms: Lactobacillus plantarum 299v
Drug: Placebo comparator — Micro-crystalline cellulose powder, identical taste, texture and appearance
  Arms: Crytalline cellulose powder
Other: Run in period — Run -in period of one to two weeks. No treatment. Treatment started at baseline following randomization to either L.plantarum 299v or placebo
  Other Names: Run in period to baseline
  Arms: Crytalline cellulose powder; Lactobacillus plantarum 299v
Other: Wash - out period — Wash - out period following treatment phase of eight weeks
  Other Names: Wash - out following treatment phase of eight weeks
  Arms: Crytalline cellulose powder; Lactobacillus plantarum 299v

SUMMARY:
In patients with IBS, will supplementation with a probiotic demonstrate symptomatic efficacy and will the probiotic influence gut microflora and thus improve clinical outcomes, as compared to no intervention.

DETAILED DESCRIPTION:
Conduct a study on nutrient intakes gastrointestinal microbiota and the effect of a probiotic, Lactobacillus plantarum 299v in irritable bowel syndrome patients.

ELIGIBILITY:
Inclusion Criteria:

* fulfillment of the Rome II criteria for IBS,
* availability of at least one colonoscopy within the last three years,
* aged 18 or older at the time of screening,
* provision of written informed consent,
* commitment of availability throughout the 12 week study period.

Exclusion Criteria:

* major abdominal surgery in the past other than other than appendectomy, caesarean section, tubal laparoscopic cholecystectomy, abdominal wall hernia repair or/and hysterectomy,
* current use of antibiotics,
* history of organic intestinal disease,
* pregnant or breastfeeding mothers,
* chronic infectious disease like HIV or tuberculosis, and
* unable to understand English or Afrikaans.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2011-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl Stevenson, M.Sc, Principal Investigator — Univeristy of Stellenbosch
Locations (1):
- Netcare Greenacres Hospital, Port Elizabeth, Eastern Cape, South Africa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at a private gastroenterology clinic in Port Elizabeth, South Africa between January 2011- June 2013,
Pre-assignment Details: Run-in phase of 1-2 weeks, then an 8 week treatment phase followed by a 2 week wash out period.
Groups:
- Lactobacillus Plantarum 299v: Treatment Lactobacillus plantarum 299v
- Placebo: Controls Crytalline cellulose powder
Period: Overall Study
Arm/Group | Lactobacillus Plantarum 299v | Placebo
Started | 54 | 27
Completed | 40 | 25
Not Completed | 14 | 2
Not completed — Protocol Violation | 5 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 5 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Worsening of symptoms | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Plantarum 299v | Placebo | Total
Number analyzed (Participants) | 54 | 27 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.15 (13.48) | 47.27 (12.15) | 47.86 (13.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 27 | 79
  Male | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  South Africa | 54 | 27 | 81
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.83 (7.12) | 28.88 (7.74) | 28.85 (7.32)
Duration of IBS (years) [Mean (Standard Deviation); unit: years] | 9.58 (10.32) | 10.05 (9.36) | 9.74 (10)

OUTCOME MEASURES:

1. Primary Outcome: A Change in Abdominal Pain Severity
Description: The clinical severity of the IBS symptoms (pain and distension) was evaluated by the Francis Severity Score questionnaire (Francis 1997). The questionnaire is a validated tools for use in IBS. The severity score contained five questions, each given a value from 0 (no symptoms) to 100 (most severe) for measuring the severity and frequency of abdominal pain. The sum of scores of these questions was considered the severity score, with a maximum possible score of 500
Time Frame: Total trial period 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lactobacillus Plantarum 299v | Placebo
Number analyzed (Participants) | 40 | 25
units on a scale
  Baseline | 259.66 (106.90) | 256.04 (104.27)
  End of treatment at week 8 | 199.13 (119.70) | 201.98 (97.44)
  Change | 60.53 (12.8) | 54.06 (6.83)
Statistical Analysis 1: Comparison: Lactobacillus Plantarum 299v vs Placebo; An intention-to -treat (ITT) analysis was performed on all patients who underwent randomization (n = 81). The results of the ITT analysis are presented. Changes in Severity Score was examined using the mixed model for analysis of variance to account for missing data. This model used group (treatment vs control) & time as factors; Test type: Non-Inferiority or Equivalence — To determine an effect size of 0.64 with 80% power, a sample size of 27 for each group (D-IBS, C-IBS and controls), with a type 1 error of 5% using a two sided test was sufficient. Sample size based on expected behaviour of primary outcome measure. The minimally clinically important difference based on the primary outcome measure with the instrument used was 50 points; p < 0.05, Mixed Models Analysis

ADVERSE EVENTS:
Arm/Group | Lactobacillus Plantarum 299v | Placebo
Serious Adverse Events (participants affected / at risk) | 1/54 | 0/27
Other Adverse Events (participants affected / at risk) | 0/54 | 0/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lactobacillus Plantarum 299v (N=54) | Placebo (N=27)
Severe rash (Reproductive system and breast disorders) | 1 | 0 — Severe rash unrelated to test product

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No